CLINICAL TRIAL: NCT00115687
Title: Nicotine Replacement Treatment for Pregnant Smokers
Brief Title: Nicotine Replacement Treatment for Pregnant Smokers - 1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy rates did not show large enough differences between treatments
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Cheryl Oncken, MD, MPH, University of Connecticut School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-15167-1; R01-15167-1; DPMCDA; NCT00064948 (obsolete NCT alias)
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2010-05

CONDITIONS: Tobacco Use Disorder
Keywords: nicotine addiction
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Placebo Comparator): placebo
  Interventions: Drug: placebo
- B (Experimental): 2 mg nicotine gum
  Interventions: Drug: 2 mg nicotine polacrilex

INTERVENTIONS:
Drug: placebo
  Arms: A
Drug: 2 mg nicotine polacrilex
  Arms: B

SUMMARY:
Smoking during pregnancy is an important modifiable cause of poor pregnancy outcomes. Even with augmented behavioral interventions, smoking cessation rates in pregnancy trials rarely exceed 20%. These low quit rates may be due to inadequate treatment of the physical dependence on nicotine. Indeed, medications, which may help to reduce nicotine withdrawal symptoms, are a first-line treatment for smoking treatment in non-pregnant smokers. However, little information is available on the safety or efficacy of medications to treat pregnant smokers.

The purpose of this trial is to evaluate the safety and effectiveness of 2 mg nicotine gum in promoting smoking cessation during pregnancy. The design is a randomized, placebo controlled trial where subjects are randomized to nicotine gum (6 weeks ad libitum use followed by a 6 week taper) or a matching placebo. Women who are doing well at the end of the trial will also be offered gum post-partum for relapse prevention.

DETAILED DESCRIPTION:
This proposal will examine the utility of one first-line medication, nicotine gum, as an aid to smoking cessation during pregnancy.

The specific aims are:

* (1) To compare smoking cessation rates and smoking reduction among pregnant smokers who are randomized to receive nicotine gum (2 mg dose) or a matching placebo;
* (2) To compare nicotine gum versus placebo on surrogate measures of maternal and fetal safety (i.e., overall nicotine and tobacco exposure at 6 weeks after the quit date and at 32-34 weeks gestation) and birth weight at the time of delivery;
* (3) To examine which subjects benefit the most from the use of nicotine gum for smoking cessation during pregnancy.

Subjects will be recruited from prenatal clinics that serve primarily a low-income, minority population. Two hundred sixty-eight pregnant smokers will be randomly assigned to receive smoking cessation behavioral counseling and either a 6-week course of mint flavored placebo or nicotine gum, followed by 6 weeks of decreasing doses. Maternal blood for genotyping will be obtained at study entry. Primary outcome measures will be 7-day point prevalence of cigarette abstinence, number of cigarettes smoked per day, urinary cotinine concentrations, and measures of tobacco exposure (i.e., carbon monoxide in exhaled air and urine anabasine and anatabine) at 6 weeks after the quit date and at 32-34 weeks gestation, and infant birth weight. We hypothesize that:

* (1) Pregnant smokers who are randomized to nicotine gum will have double the quit rates and will reduce their smoking to a greater degree than subjects randomized to placebo;
* (2) Nicotine gum compared to placebo will reduce maternal levels of tobacco-exposure markers and increase birth weights in the offspring;
* (3) The odds of cigarette abstinence will be increased primarily in subjects who smoke at least 15 cigarettes per day.

ELIGIBILITY:
Inclusion Criteria:

* Patient's gestational age is 26 weeks or less.
* Patient is at least 16 years of age.
* Patient is able to speak English or Spanish.
* Patient intends to carry to term.
* Patient has stable residence.
* Patient has smoked five or more cigarettes everyday for the past seven days.

Exclusion Criteria:

* Evidence that the patient is pregnant with a fetus with a known congenital abnormality.
* Unstable medical problems (i.e., hyperthyroidism, temporomandibular joint disorder, pre-eclampsia, threatened abortion, hyperemesis gravidarum)
* Multiple Gestation
* Unstable psychiatric disorder
* Current drug or alcohol abuse or dependence

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Actual)
Dates: Start 2002-06; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Biochemically validated quit rates | 6 weeks after treatment, end of pregnancy

SECONDARY OUTCOMES:
tobacco exposure measurements | 6 weeks after treatment, end of pregnancy
birth weight | time of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl A Oncken, M.D., Principal Investigator — UConn Health
Locations (4):
- United States (4):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Baystate Medical Center, Springfield, Massachusetts

REFERENCES:
- [Result] Oncken C, Dornelas E, Greene J, Sankey H, Glasmann A, Feinn R, Kranzler HR. Nicotine gum for pregnant smokers: a randomized controlled trial. Obstet Gynecol. 2008 Oct;112(4):859-67. doi: 10.1097/AOG.0b013e318187e1ec. PMID 18827129